CLINICAL TRIAL: NCT02032485
Title: Feasibility Study of the (Intravenously Injected) Indocyanine Green (ICG) Imaging of Tumoral Implants in Patients With Peritoneal Carcinomatosis From Colorectal Cancer
Brief Title: Near-Infrared Imaging of Peritoneal Carcinomatosis From Colorectal Cancer
Acronym: OC-AP-ICG-IV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-000653-42
Record Dates: First submitted 2013-11-20; First posted 2014-01-10 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-07

CONDITIONS: Colorectal Cancer; Peritoneal Carcinomatosis
Keywords: colorectal cancer; Indocyanine Green; visualization of peritoneal metastases
MeSH Terms: conditions — Colorectal Neoplasms; Peritoneal Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Indocyanine Green (Experimental): Intravenous injection of 0.25 mg/kg Indocyanine Green in patients with peritoneal carcinomatosis from colorectal cancer before the surgery
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — An iv injection will be performed for the colorectal cancer patient before the operation.
  Other Names: ICG

SUMMARY:
The purpose of this study is to determine if Near-Infrared fluorescence imaging is an effective approach to detect the colorectal tumoral tissues and peritoneal implants in colorectal cancer patients.

DETAILED DESCRIPTION:
Primary objective

Evaluation of the ability of NIR imaging using ICG to demonstrate (the gross tumoral mass and/or) peritoneal metastatic " implants " in patients operated for peritoneal carcinomatosis from colorectal carcinoma

Secondary objective:

Definition of the histological distribution (in the vessels, in the extravascular spaces, in specific cells) of IV injected ICG in the normal and pathological tissues (and, if any is demonstrated per-operatively, a) in the nodes of these patients found fluorescent and removed and/or b) at the level of the fluorescent foci observed at the level of the hepatic surfaces)

Methodology:

The day before the operation:

ICG 0.125 mg/kg will be given as an iv injection the day before the operation.

In the operating room:

When the patient will be operated, the surgeons will (under "conventional" video control) search and establish as usual the presence (of "gross" tumoral mass and) of metastatic deposits at the level of the peritoneal surfaces. NIR imaging will be acquired during these manoeuvers and, if detected, fluorescent structures and/or foci will be anatomically defined by the surgeons.

If ("gross" tumoral mass and/or) metastatic deposits are seen fluorescent, the operation will be then continued as usual but each anatomical piece will be controlled "ex vivo" for its fluorescent character or not. All fluorescent foci on these anatomical pieces will be identified as such by a mark and/or by a "suture".

If ("gross" tumoral mass and/or) metastatic deposits are not seen fluorescent, ICG 0.125 mg/kg will be given as an iv injection and the vascularization, income of the ICG in the tumoral implants (judged by the surgeon the most representative of the patient's status) will be dynamically studied using the PDE camera during the 10 minutes following the IV injection.

If no hepatic metastases were pre-operatively documented, the surface of the liver will be controlled and, if superficial fluorescent foci are observed, these will be biopsied.

In the Laboratory of Pathology:

The tumoral tissues as well as -if identified- the "non identified as tumoral" fluorescent tissular foci will be processed as usual.

All the slides obtained will be analyzed using the near-infrared fluorescence microscope for the presence or the absence of (detectable) ICG and the different ICG-positive compartments (vascular spaces, interstitial spaces, normal and/or tumoral cells, macrophages,…) will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Patients (either newly diagnosed, or relapsing) with peritoneal carcinomatosis from histo-pathologically proven colorectal carcinoma who are candidate for "open" surgery,
* Informed consent form signed.

Exclusion Criteria:

* Age less than18 years old.
* Inability to give informed consent.
* History of allergy or hypersensitivity against the investigational product (its active substance or ingredients), to iodine or to shellfish.
* Apparent hyperthyroidism, autonomous thyroid adenoma, unifocal, multifocal or disseminated autonomy of the thyroid gland.
* Documented coronary disease.
* Advanced renal impairment (creatinine > 1,5mg/dl).
* During the 2 weeks before the enrolment, concurrent medication which reduces or increases the extinction of ICG (i.e. anticonvulsants, haloperidol and Heparin).
* Pregnancy, breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
fluorescence intensity of tumoral and healthy tissues after IV injection of ICG to patients with peritoneal carcinomatosis from colorectal origin. | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Liberale, MD, Principal Investigator — Surgeon in Jules Bordet Institute
Locations (1):
- Institut Jules Bordet, Brussels, Brussels Capital, Belgium